CLINICAL TRIAL: NCT03464071
Title: Biomarkers of Lung Injury in the Hyperinflation Maneuver in the Mechanical Ventilator Versus Manual Hyperinflation in Septic Patients: Randomized Clinical Trial
Brief Title: Biomarkers of Lung Injury in Hyperinflation in the Mechanical Ventilator Versus Manual Hyperinflation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 170580
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-03

CONDITIONS: Sepsis
Keywords: sepsis; biomarkers; lung injury
MeSH Terms: conditions — Sepsis; Lung Injury | interventions — Ventilators, Mechanical

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group HVM (Experimental): When randomized to the Hyperinflation with mechanical ventilator (HVM) group, there will be an increase in initial positive inspiratory pressure until reaching a peak pressure of 40 cmH2O and PEEP equal to 7 cmH2O
  Interventions: Device: Hyperinflation with mechanical ventilator
- Group HM (Experimental): When randomized to the Manual hyperinflation (HM) group, the manual resuscitation bag will be connected to the oxygen system at five liters per minute. The participant will be disconnected from the ventilator and then initiate a slow inspiration with inspiratory pause followed by abrupt expiration, totaling twelve (12) cycles / minute.
  Interventions: Device: Manual hyperinflation

INTERVENTIONS:
Device: Hyperinflation with mechanical ventilator — increase in initial positive inspiratory pressure until reaching a peak pressure of 40 cmH2O and PEEP equal to 7 cmH2O
  Arms: Group HVM
Device: Manual hyperinflation — the manual resuscitation bag will be connected to the oxygen system at five liters per minute. The participant will be disconnected from the ventilator and then initiate a slow inspiration with inspiratory pause followed by abrupt expiration, totaling twelve (12) cycles / minute.
  Arms: Group HM

SUMMARY:
Due to the failure of the respiratory system, many patients admitted to the Intensive Care Units (ICUs) require the institution of invasive mechanical ventilation (MV), aiming at maintaining gas exchange, reversing respiratory muscle fatigue, among other benefits. However, an artificial airway installation may be harmful because of its deleterious capacity to the mucociliary clearance mechanism, predisposing to the accumulation of secretions and consequent respiratory infections. Physiotherapy in patients critical for the purpose of preventing and treating these respiratory complications. In this way, they are techniques that aim at a reexpansion and removal of airborne secretions. An application of manual hyperinflation with the Ambú (HM), applied through compression of the resuscitator (Ambu), an application of hypertension for the use of energy, pulmonary volume. Similar to the goal of manual hyperinflation, a hyperinflation maneuver without mechanical ventilator (HVM) is also widely used and has been shown to be effective. A maneuvering visa re-expansion of collapsed lung areas and increased peak expiratory flow, resulting in the mobilization of secretions. It is known that these techniques can cause deleterious effects to the lungs due to the high volumes administered and the variation in airway depression, predisposing to barotrauma and volutrauma, increasing the lung permeability and consequent pulmonary edema. There may also be a more subtle form of injury, such as a release of lung mediators, initiating a process of local inflammation. This biological response is called biotrauma, and if these mediators translocate into the systemic circulation, it can lead to dysfunction and death. The aim of the present study was to evaluate the biomarkers of pulmonary lesion in the hyperinflation maneuver with mechanical ventilator versus manual hyperinflation with environments in sudden patients under mechanical ventilation.

DETAILED DESCRIPTION:
This study aims to evaluate the biomarkers of lung injury in the hyperinflation maneuver with mechanical ventilator versus manual hyperinflation with ambu in septic patients under mechanical ventilation through changes in the cellular levels of interleukin 8 (IL-8) and receptor for advanced glycation end products (RAGE). As specific objectives, compare the variables of ventilatory mechanics (dynamic compliance, static complacency, frequency airway resistance) and hemodynamic parameters (systolic blood pressure, diastolic blood pressure, mean arterial pressure and heart rate) before and after each maneuver and between groups. It is characterized as a randomized clinical trial. The binary randomization of the groups will be performed using the electronic application Bracket RTSM (version 2.0.0, Bracket Global), and will be performed by a blind researcher to the groups evaluated. After the eligibility criteria, the selected patients will be randomized and divided into two groups : Hyperinflation group with mechanical ventilator (HVM) and manual hyperinflation group (HM). Triage will be carried out daily in order to detect patients eligible to apply the study through communication with the local multiprofessional team. Once patients are eligible according to the inclusion and exclusion criteria, randomization will be performed to determine the techniques to be employed. Prior to the application of each technique, all patients will be placed in the dorsal decubitus (DD) with the head elevated at 30 degrees and will be aspirated by the nursing team once with probe number nº 14 and with a vacuum of -40cmH2O. Five minutes later, a 4.5 mL blood sample from the study participant for analysis of lung injury biomarkers (IL-8 and RAGE) will be collected in an EDTA tube. Blood samples will be sent to the Molecular and Protein Analysis Unit (UAMP) of the HCPA Experimental Research Center (CPE) in a box cooled by a blind collaborator who is not part of the study and will be stored at -80ºC. The biomarkers will be tested in duplicates through the plasma of the sample collected using the Luminex Human Magnetic Assay kit (R & DSystems, Minneapolis, MN). The results will be transcribed to the datasheet. A period of five minutes will be waited for the start of the initial technique chosen by randomization. When drawn to the HVM group, there will be an increase in initial positive inspiratory pressure until reaching a peak pressure of 40 cmH2O and PEEP equal to 7 cmH2O. During the application of this technique VC will increase significantly in most patients, which may cause and / or increase Auto-PEEP. In order to minimize and / or extinguish this adverse effect the RF should be reduced to allow exhalation. When drawn to the HM group, the manual resuscitation bag will be connected to the oxygen system at five liters per minute. The participant will be disconnected from the ventilator and then initiate a slow inspiration with inspiratory pause followed by abrupt expiration, totaling twelve (12) cycles / minute. Data will be collected on ventilatory mechanics (dynamic compliance, expiratory tidal volume, respiratory rate, peak pressure, plateau pressure, airway resistance) from the ventilator used in the SERVO-s® institution and hemodynamic parameters (systolic blood pressure, diastolic blood pressure, mean arterial pressure and heart rate) in the hemodynamic monitoring device MP60® before and after the application of each technique, and the data will be recorded on an evaluation form. After each maneuver, a period of three hours will be waiting and then a blood sample will be collected again from the patient for the analysis of lung injury biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the ICPA ICU who have a minimum of 24 hours under mechanical ventilation, coupled to the orotracheal tube (TOT) or tracheostomy (TQT) in pressure-controlled ventilation (PCV) or volume-controlled ventilation (VCV) .
* Hemodynamically stable patients with mean arterial pressure equal to or greater than 60 mmHg with Noradrenaline doses of less than 0.5 μg / kg / minute.
* Septic patients.

Exclusion Criteria:

* Patients with contraindications to increased positive pressure (non-drained pneumothorax and hemothorax, subcutaneous emphysema).
* Patients with a diagnosis of adult respiratory distress syndrome (ARDS).
* Neurosurgical patients who are under intracranial pressure monitoring (ICP);
* Patients with Peak inspiratory pressure (PIP) = 40 cmH2O and / or PEEP> 10 cmH2O.
* Post-surgical patients
* Patients submitted to extracorporeal circulation (ECC)
* Chronic renal patients
* Patients without relatives.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-09-10 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Interleukin 8 (IL-8) | variation in 3 hours
  A sample of 4.5 mL of blood from the study participant for analysis of lung injury biomarkers will be collected in an EDTA tube and then analyzed using the Luminex Human Magnetic Assay kit
Receptor for advanced glycation end products (RAGE) | variation in 3 hours
  A sample of 4.5 mL of blood from the study participant for analysis of lung injury biomarkers will be collected in an EDTA tube and then analyzed using the Luminex Human Magnetic Assay kit

SECONDARY OUTCOMES:
Systolic blood pressure | variation in 3 hours
  will be verified through the Philips MP60® hemodynamic monitoring device
Diastolic blood pressure | variation in 3 hours
  will be verified through the Philips MP60® hemodynamic monitoring device
Heart rate | variation in 3 hours
  will be verified through the Philips MP60® hemodynamic monitoring device
Mean arterial pressure | variation in 3 hours
  will be verified through the Philips MP60® hemodynamic monitoring device
Respiratory rate | variation in 3 hours
  value obtained from the ventilator used in the institution SERVO-s®
Dynamic compliance (cdyn) | variation in 3 hours
  value obtained from the ventilator used in the institution SERVO-s®
Static compliance (cst) | variation in 3 hours
  value obtained from the ventilator used in the institution SERVO-s®
Peak inspiratory pressure (PIP) | variation in 3 hours
  value obtained from the ventilator used in the institution SERVO-s®
Plateau pressure (PP) | variation in 3 hours
  value obtained from the ventilator used in the institution SERVO-s®
Airway resistance (Raw) | variation in 3 hours
  value obtained from the ventilator used in the institution SERVO-s®

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Regina Rios Vieira, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil